CLINICAL TRIAL: NCT01494779
Title: Evaluation of Pharmacokinetic and Pharmacodynamic Parameters of Somatropin Produced by Laboratory Blausiegel Indústria e Comércio Ltda., Compared to Saizen® From Laboratory Merck Serono S.A.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SOMBLA0911; Version 1
Record Dates: First submitted 2011-11-28; First posted 2011-12-19 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: GH Deficiency (GHD); Growth Retardation
Keywords: children
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

ARMS (2):
- Somatropin Test (Experimental): Somatropin of Blausiegel Indústria e Comércio Ltda.
  Interventions: Drug: Somatropin
- Saizen (Active Comparator): Somatropin of Merck Serono
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — single subcutaneous dose of 5mg
  Arms: Somatropin Test
Drug: Somatropin — single subcutaneous dose of 5mg
  Arms: Saizen

SUMMARY:
The primary objective of this study is to compare the pharmacokinetic and pharmacodynamic effect between two preparations of somatropin (T and C) after a single administration of 5 mg in healthy subjects by altering serum somatropin pharmacokinetic parameters (AUC0-24h, AUC0-inf, Cmax, Tmax and T1 / 2) and pharmacodynamic (measurement of serum levels of IGF-1 presented by the concentration-time profile, AUC 0-24h and AUC0-inf.).

DETAILED DESCRIPTION:
Secondly, the investigators will observe the clinical safety and tolerability after single dose administration in subjects, by comparing clinical parameters and the incidence of adverse events between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Research subjects who agree with all study procedures, sign and date, of their own free will, the IC;
2. Research subjects were male, aged between 18 and 32 years;
3. Research subjects with body mass index greater than or equal to 20 and less than or equal to 25;
4. Considered healthy subjects, both clinical and laboratory.

Exclusion Criteria:

1. Have donated or lost 450 mL or more blood in the 6 months preceding the study;
2. Having participated in any experimental study or have taken any experimental drug in the 12 months preceding the start of the study;
3. Having made use of regular medication less than two weeks to interfere with the pharmacokinetics / pharmacodynamics of the drug under study, such as glucocorticoids, anabolic steroids, androgens, estrogens and thyroid hormones;
4. Present history of alcohol abuse, drug or drugs;
5. Have a history of liver disease, renal, pulmonary, gastrointestinal, hematologic, or psychiatric;
6. Have made previous use of somatropin;
7. Make use of energy supplements and / or be frequent consumers of soy products (eg replacement of animal milk for soy milk).

Ages: 18 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be based in the investigation of pharmacokinetics and pharmacodynamics of somatropin in research subjects after administration of single dose, sc, of the drug. | PK: 0, 1, 2, 3, 3:30, 4, 4:30, 5, 6, 9, 12, 15, 18, 24 hours. PD: 0, 6, 12, 24 hours.
  Pharmacokinetic evaluation will be based on data obtained from the average dosage of somatropin plasma. Thus, the time of collection facilities provide the pharmacokinetic parameters AUC0-24h, AUC0-inf, Cmax, Tmax and T1 / 2, which will be compared between the two formulations.
  The quantification of serum somatropin kit will be performed by ELISA validated using human serum as a biological matrix.
  The evaluation of the pharmacodynamics will be performed by quantifying serum levels of IGF-1 presented by the concentration-time profile, AUC 0-24h and AUC0-inf.

SECONDARY OUTCOMES:
After administration of the drug will be evaluated for safety and tolerability of the drug through the presence of hematoma, pain, itching and local redness, as well as the incidence of adverse events directly related to somatropin. | 15 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil